CLINICAL TRIAL: NCT02104596
Title: Intraarticular Xylitol Injections for Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, KANDEL, Orthopedic Surgeon, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Xylitol- HMO-CTIL
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Xylitol injection (Experimental): Intraarticular injection of Xylitol
  Interventions: Device: Xylitol
- Control (Placebo Comparator)

INTERVENTIONS:
Device: Xylitol
  Arms: Xylitol injection

SUMMARY:
Hypothesis: Intraarticular injections of isotonic Xylitol solution will improve pain in patients with knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Age over 45
* Tibiofemoral osteoarthritis
* OA stage 2-3 on xray
* Pain VAS > 40mm
* No NSAIDs for 3 weeks
* No analgetics for 38 hours

Exclusion Criteria:

* Pain VAS > 80mm
* Pain VAS in contralateral knee > 40mm
* Inflammatory arthritis
* Severe effusion
* Posttraumatic osteoarthritis
* Unstable knee
* Isolated patellofemoral disease
* Paracetamol hypersensitivity

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Pain - visual analogue scale | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel